CLINICAL TRIAL: NCT03106038
Title: A Phase I/IIa Dose-escalation Study to Evaluate the Use of an Investigational Imaging Agent for the Detection of Urologic Anatomy Via Near Infrared Fluorescence Imaging in the Setting of Minimally Invasive Surgery
Brief Title: Dose-escalation Study of a Contrast Agent for Delineation of Urological Anatomy in Minimally Invasive Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Li-Cor, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: LICOR-10417-01
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Intraoperative Ureter Injury
Keywords: contrast agent; ureter imaging; intraoperative monitoring; intraoperative procedures; near infrared fluorescence; minimally invasive
MeSH Terms: interventions — Injections; IRDye 800BK

STUDY DESIGN:
Intervention Model Description: beginning at the estimated target dose, the dosage was increased and decreased to confirm the near-optimal dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nerindocianine for Injection (Experimental): One Arm: Nerindocianine for Injection (Initial dosing cohort: 0.06 mg/kg body weight); solution, intravenous, one time administration during surgery. the study has only one arm.
  Interventions: Drug: Nerindocianine for Injection

INTERVENTIONS:
Drug: Nerindocianine for Injection — Procedure: routine minimally invasive pelvic surgery.
  Other Names: IRDye 800BK

SUMMARY:
The purpose of this clinical trial is to study the safety and efficacy of an investigational imaging agent for delineation/visualization of urologic anatomy in the setting of minimally invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to the initiation of study procedures
* Are > 18 years of age
* Women consented to undergo standard of care minimally invasive pelvic surgery (traditional laparoscopy and robotic surgery)
* Women who are expected to be admitted to the hospital following surgery for at least 24 hours

Exclusion Criteria:

* Are unwilling or unable to provide informed consent.
* Are unwilling or unable to comply with the requirements of the protocol.
* History of prior urologic surgery.
* History of prior pelvic surgery.
* History of known retroperitoneal fibrosis.
* Have any of the following screening laboratory values:

  * Hemoglobin ≤ 8.0 g/dL;
  * Absolute neutrophil count (ANC) ≤ 1500/μL;
  * Platelet count ≤ 100,000/μL;
  * Serum creatinine ≥ 1.5 x the institutional upper limit of normal (IULN) creatinine;
  * Serum bilirubin ≥ 1.5 x IULN;
  * Aspartate transaminase (AST or serum glutamic oxaloacetic transaminase, SGOT) ≥ 2x IULN;• Alanine transaminase (ALT or serum glutamate pyruvate transaminase, SGPT) ≥ 2 x IULN.
* Females who are pregnant, lactating, or breastfeeding;
* Any other condition that, in the Investigator's judgment, would potentially compromise the study compliance or the ability to evaluate safety or efficacy.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 30 days
  Incidence of Treatment-Emergent Serious Adverse Events and/or Treatment-Emergent Adverse Events
Dose response | 10 minutes through 90 minutes post administration
  Dose response based on the composite assessment of the anatomy and laterality for detection of pelvic ureter in women undergoing minimally invasive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H. Kim, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Women & Infants Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh WK, Johnson JL, Elliott E, Boone JD, Leath CA 3rd, Kovar JL, Kim KH. Fluorescence Imaging of the Ureter in Minimally Invasive Pelvic Surgery. J Minim Invasive Gynecol. 2021 Feb;28(2):332-341.e14. doi: 10.1016/j.jmig.2020.06.022. Epub 2020 Jun 29. PMID 32615331